CLINICAL TRIAL: NCT04741191
Title: Effects of Cycle Ergometer Training on Heart Rate Recovery and Mind Fullness in NYHA Class I, II Heart Failure Patients
Brief Title: Cycle Ergometer Training and Heart Failure on Heart Rate Recovery and Mind Fullness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/00784 Irfan ullah
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure NYHA Class I; Heart Failure NYHA Class II
Keywords: Cycle ergometer; Heart rate recovery; Mindfulness; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycle ergometer training (Experimental): Hospital-based ergometer cycling for 20 minutes (Including warm-up and cooldown)
  Interventions: Other: Cycle ergometer training
- Conventional therapy (Active Comparator): Patient education and counseling, In bed activities, Ambulation
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Cycle ergometer training — Hospital-based ergometer cycling for 20 minutes (Including warm-up and cooldown), 3x/week on alternate days for 6 weeks at 40-60% of VO2max.
  Arms: Cycle ergometer training
Other: Conventional therapy — In bed activities (Active ankle and hand pumping exercise* 15 Rep* BD AROMS of extremities* 15 Rep* BD, Deep breathing exercises* 15 Rep* BD, Ambulation (walk 10-15 minutes below fatigue and onset of symptoms level* BD) for 6 weeks.
  Arms: Conventional therapy

SUMMARY:
To evaluate the effects of cycle ergometer training on heart rate recovery in Newyork Heart Association (NYHA) class I and II heart patients. To evaluate the effects of cycle ergometer training on mind fullness in NYHA class I and II heart patients. Previous studies were designed to target only cardiac functions and no psychological aspect was studied so this study cover this aspect as well so from the outcomes of this study we can determine both psychological satisfaction and cardiac function as well.

DETAILED DESCRIPTION:
A review stated that "clinical and experimental data shows that physical training is an important aspect in the management of chronic heart failure patients. Also, it stated that physical exercise training plays an important role to modulate peripheral immune responses if congestive heart failure (CHF) patients show high pro-inflammatory cytokines, soluble cellular adhesion molecules, which further resulted in an improvement in exercise capacity in CHF patients.

Heart rate recovery (HRR) improved in patients who were enrolled in the cardiac rehabilitation stage 2 program while similar outcomes were not noted among the control group. It was concluded that cardiac rehabilitation exercise program improves heart rate recovery. Also, HRR may be used in a cardiac rehabilitation program to recognize high risk factors and also useful in evaluating the outcomes.

a systematic review about the effects of exercise training in patients with CHF was published who concluded that short-term physical exercise training in selected subgroups of patients with CHF, has physiological benefits and positive effects on quality of life.

A meta-analysis by the Collaborative Group concluded that there is no evidence that supervised medical training programs for patients with CHF are dangerous and indeed there is clear evidence of an overall reduction in mortality. The authors did not perform a quantitative analysis on the outcome of cardiac performance, exercise capacity, or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Vitally stable Patients with HF 6-8 weeks post-discharge from the hospital
* NYHA class I, II
* EF: 25-40%

Exclusion Criteria:

* Arrhythmias /Regular Pvc/Permanent pacemaker/Tpm
* Any systematic disease /infections
* Uncontrolled DM/HTN
* Unable to perform the 6-min walk test

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Heart rate recovery | 6 weeks
  Changes from the baseline will be measured after every intervention session. Heart rate recovery is normally measured at 1, 2 or 3-minute intervals, with 1-minute HRR being the one that is most commonly used. For example, if your heart rate is 170 beats per minute when you finish working out, and then it drops to 150 bpm a minute later, your HRR is 20 bpm.

SECONDARY OUTCOMES:
Mindfulness | 6 weeks
  A mental state achieved by focusing one's awareness on the present moment, while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations, used as a therapeutic technique. It is measured through a scale that assesses characteristics of mindfulness which consist of 15-items. It assesses the present situation, perception or attention of mind, to observe what is going to happen, and sensitive awareness of what is occurring in the present.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital,, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu CY, Hsieh PL, Hsiao SF, Chien MY. Effects of Exercise Training on Autonomic Function in Chronic Heart Failure: Systematic Review. Biomed Res Int. 2015;2015:591708. doi: 10.1155/2015/591708. Epub 2015 Oct 12. PMID 26543861
- [Background] Yaylali YT, Findikoglu G, Yurtdas M, Konukcu S, Senol H. The effects of baseline heart rate recovery normality and exercise training protocol on heart rate recovery in patients with heart failure. Anatol J Cardiol. 2015 Sep;15(9):727-34. doi: 10.5152/akd.2014.5710. Epub 2014 Oct 15. PMID 25592094
- [Background] van Tol BA, Huijsmans RJ, Kroon DW, Schothorst M, Kwakkel G. Effects of exercise training on cardiac performance, exercise capacity and quality of life in patients with heart failure: a meta-analysis. Eur J Heart Fail. 2006 Dec;8(8):841-50. doi: 10.1016/j.ejheart.2006.02.013. Epub 2006 May 18. PMID 16713337
- [Background] Piepoli MF, Davos C, Francis DP, Coats AJ; ExTraMATCH Collaborative. Exercise training meta-analysis of trials in patients with chronic heart failure (ExTraMATCH). BMJ. 2004 Jan 24;328(7433):189. doi: 10.1136/bmj.37938.645220.EE. Epub 2004 Jan 16. PMID 14729656